CLINICAL TRIAL: NCT02606357
Title: Treatment Initiation With Basal Insulin in Uncontrolled Type 2 Diabetes Patients on Oral Anti-Diabetic Agent (OAD) in Jordan
Brief Title: Treatment of Type 2 Diabetes With Long Acting Basal Insulin in Jordan
Acronym: NEWLAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LANTUL07225; U1111-1172-1002 (Other: UTN)
Record Dates: First submitted 2015-11-13; First posted 2015-11-17 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HOE901 (Experimental): HOE901 administered subcutaneously once a day in the evening, at dinner, or at bedtime with titration based on FPG levels
  Interventions: Drug: INSULIN GLARGINE

INTERVENTIONS:
Drug: INSULIN GLARGINE — Pharmaceutical form:Solution
  Route of administration: Subcutaneous
  Other Names: HOE901

SUMMARY:
Primary Objective:

-To assess the change in glycosylated hemoglobin (HbA1c) in uncontrolled Type 2 diabetes patients on OAD agent in Jordan after 6 months of treatment with basal insulin (Insulin glargine).

Secondary Objectives:

* To evaluate the percentage of patients achieving target of HbA1c ˂7%.
* To evaluate the change in fasting plasma glucose (FPG).
* To assess the following safety criteria: hypoglycemic events, body weight changes, and overall safety.
* Describe the titration process: changes in glargine insulin dose at 3 months and 6 months, changes in the titration doses used (if any), and time to reach control.

DETAILED DESCRIPTION:
The total duration of study period per patient is up to 6 months.

ELIGIBILITY:
Inclusion criteria :

* Patient ≥ 18 years old.
* Male or Female.
* Type 2 diabetes patients.
* Uncontrolled with previous therapy (HbA1c >7%), evident in HbA1c test within the last 1 month before study entry.
* Insulin naïve patients: any patient uncontrolled after one or a maximum of two lines of therapy including: monotherapy (Metformin alone or any other Oral Anti-Diabetic agent (OAD) if contraindicated or intolerance) and/or dual therapy (any OAD combination), at maximum tolerated dose in the last 3 months.
* Signed informed consent.
* Signed informed consent.

Exclusion criteria:

* Patient not willing or not able to perform self-monitoring blood glucose.
* Patient not willing or not able to self-titrate insulin glargine under physician's guidance.
* Patient not suitable for participation according to what is specified in the approved Summary of Product's Characteristics or according to medical or clinical conditions, as judged by the Investigator.
* History of impaired hepatic function defined as alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) greater than three times the upper limit of normal, evident in testing done in the last 3 months.
* History of impaired renal function defined as serum creatinine >135 μmol/L (>1.525 mg/dL)in men and >110 μmol/L (>1.243 mg/dL) in women, evident in testing done in the last 3 months.
* Pregnant or lactating women (women of childbearing potential must have a negative pregnancy test at study entry and a medically approved contraception method at physician's discretion).
* Treatment with systemic corticosteroid within 3 months prior to study entry.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2015-11-22 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | Baseline, 6 months

SECONDARY OUTCOMES:
- Percentage of patients achieving target of HbA1c <7% | 6 months
- Change from baseline in fasting plasma glucose values | Baseline, 3 months, and 6 months
- Percentage of patients with hypoglycemic events | Baseline, 6 months
- Change from baseline in body weight | Baseline, 3 months and 6 months
- Number of patients with adverse events | Baseline, 6 months
- Change in dose of insulin glargine | 3 months and 6 months
- Change in the titration doses used (if any) | 6 months
- Time to reach control | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- JORDAN, Jordan, Jordan